CLINICAL TRIAL: NCT04161898
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Upadacitinib in Subjects With Takayasu Arteritis (SELECT-Takayasu)
Brief Title: A Study to Evaluate the Efficacy and Safety of Upadacitinib in Participants With Takayasu Arteritis (TAK)
Acronym: SELECT-TAK
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M19-052
Record Dates: First submitted 2019-11-12; First posted 2019-11-13 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Takayasu Arteritis (TAK)
Keywords: Takayasu Arteritis (TAK); Upadacitinib; Placebo; Corticosteroid; Prednisolone
MeSH Terms: conditions — Takayasu Arteritis | interventions — upadacitinib; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1: Upadacitinib (Experimental): Participants will be administered updadacitinib once daily (QD) along with prednisolone.
  Interventions: Drug: Upadacitinib; Drug: Prednisolone
- Arm 2: Placebo for Upadacitinib (Experimental): Participants will be administered placebo once daily (QD) along with prednisolone.
  Interventions: Drug: Upadacitinib; Drug: Placebo for Upadacitinib; Drug: Prednisolone

INTERVENTIONS:
Drug: Upadacitinib — Upadacitinib will be administered as oral tablet
  Other Names: ABT-494; RINVOQ
Drug: Placebo for Upadacitinib — Placebo for upadacitinib will be administered as oral tablet
  Arms: Arm 2: Placebo for Upadacitinib
Drug: Prednisolone — Prednisolone will be administered as oral tablet

SUMMARY:
The main objective of this study is to evaluate the efficacy of upadacitinib in combination with a corticosteroid taper regimen compared to placebo in combination with a corticosteroid taper regimen.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age (at least 15 years of age in Japan)
* Clinical diagnosis of TAK and fulfilling the Japanese Guidelines for Management of Vasculitis Syndrome 2017 criteria.
* Participant must have experienced a relapse of TAK within 12 weeks of Baseline despite being on treatment with oral corticosteroid.
* Participants must be in remission and on a stable corticosteroid dose prior to Baseline.

Exclusion Criteria:

* Treatment with an interleukin-6 (IL-6) inhibitor or Janus Kinase (JAK) inhibitor (including but not limited to tocilizumab, sirukumab, sarilumab, upadacitinib, tofacitinib, baricitinib, ruxolitinib, peficitinib, and filgotinib) within 4 weeks of Baseline.
* Current use of immunomodulators other than corticosteroids.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-02-04 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Time to First Relapse of Takayasu Arteritis (TAK) From Baseline through End of the Double-Blind (DB) Period | Up to occurrence of 40 events (approximately 52 months)
  Relapse of TAK is defined as the presence of signs or symptoms as judged by the investigator for at least 2 of the following categories: objective systemic symptoms, subjective systemic symptoms, elevated inflammation markers, vascular signs and symptoms, or ischemic symptoms OR where the criteria are met based on one category per protocol definition of relapse of TAK.

SECONDARY OUTCOMES:
Time to First Relapse of Takayasu Arteritis (TAK) by Kerr Criteria From Baseline through End of the DB Period | Up to occurrence of 40 events (approximately 52 months)
  Kerr criteria for relapse are defined as the presence of signs or symptoms as judged by the investigator for at least 2 of the following categories: objective or subjective systemic symptoms, elevated inflammation markers, vascular or ischemic signs and symptoms, or worsening in imaging assessment due to TAK.
Time to Worsening of Imaging Assessment Due to Takayasu Arteritis (TAK) From Baseline through End of the DB Period | Up to occurrence of 40 events (approximately 52 months)
  Imaging with computed tomography angiogram (CTA).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (48):
- Argentina (2):
  - Fundación Sanatorio Guemes /ID# 249675, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Hospital Italiano La Plata /ID# 249269, La Plata, Buenos Aires
- Brazil (6):
  - SER - Servicos Especializados em Reumatologia da Bahia /ID# 243125, Salvador, Estado de Bahia
  - CMiP - Centro Mineiro de Pesquisa Ltda - ME /ID# 242517, Juiz de Fora, Minas Gerais
  - CETI - Centro de Estudos em Terapias Inovadoras /ID# 242502, Curitiba, Paraná
  - LMK Sevicos Medicos S/S /ID# 240645, Porto Alegre, Rio Grande do Sul
  - Hospital do Rim /ID# 240380, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao /ID# 241175, São Paulo
- China (5):
  - Xuanwu Hospital Capital Medical University /ID# 248104, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital /ID# 248350, Guangzhou, Guangdong
  - Shenzhen People's Hospital /ID# 248347, Shenzhen, Guangdong
  - The First Hospital of China Medical University /ID# 248107, Shenyang, Liaoning
  - Zhongshan Hospital Fudan University /ID# 247159, Shanghai, Shanghai Municipality
- Japan (23):
  - Chiba University Hospital /ID# 214932, Chiba, Chiba
  - Ehime University Hospital /ID# 215424, Toon-shi, Ehime
  - Maebashi Red Cross Hospital /ID# 230513, Maebashi, Gunma
  - Duplicate_Hokkaido University Hospital /ID# 215066, Sapporo, Hokkaido
  - University of Tsukuba Hospital /ID# 215318, Tsukuba, Ibaraki
  - Kagawa University Hospital /ID# 214776, Kita-gun, Kagawa-ken
  - St Marianna University School Of Medicine /ID# 214535, Kawasaki-shi, Kanagawa
  - Yokohama City University Hospital /ID# 214345, Yokohama, Kanagawa
  - Duplicate_Kyoto University Hospital /ID# 215128, Kyoto, Kyoto
  - Tohoku University Hospital /ID# 214066, Sendai, Miyagi
  - Miyagi Children's Hospital /ID# 248390, Sendai, Miyagi
  - Nagano Red Cross Hospital /ID# 214537, Nagano, Nagano
  - Duplicate_Nagasaki University Hospital /ID# 215683, Nagasaki, Nagasaki
  - Okayama University Hospital /ID# 214499, Okayama, Okayama-ken
  - National Hospital Organization Osaka Minami Medical Center /ID# 228779, Kawachinagano Shi, Osaka
  - Kindai University Hospital /ID# 216491, Osakasayama-shi, Osaka
  - National Cerebral and Cardiovascular Center /ID# 214061, Suita-shi, Osaka
  - Juntendo University Hospital /ID# 214292, Bunkyo-ku, Tokyo
  - Institute of Science Tokyo Hospital /ID# 214138, Bunkyo-ku, Tokyo
  - St.Luke's International Hospital /ID# 214067, Chuo-ku, Tokyo
  - Duplicate_Keio University Hospital /ID# 214905, Shinjuku-ku, Tokyo
  - Center hospital of the National Center for Global Health and Medicine /ID# 214931, Shinjuku-ku, Tokyo
  - Duplicate_Tokyo Women's Medical University Hospital /ID# 215129, Shinjuku-ku, Tokyo
- South Korea (5):
  - Seoul National University Hospital /ID# 213844, Seoul, Seoul Teugbyeolsi
  - Hanyang University Seoul Hospital /ID# 213842, Seoul, Seoul Teugbyeolsi
  - Gangnam Severance Hospital /ID# 229543, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Marys Hospital /ID# 214566, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 215643, Seoul
- Turkey (Türkiye) (7):
  - Hacettepe University Faculty of Medicine /ID# 239845, Ankara
  - Ankara Univ Medical Faculty /ID# 240015, Ankara
  - Akdeniz University Faculty /ID# 239847, Antalya
  - Basaksehir Cam ve Sakura Sehir Hastanesi /ID# 239846, Istanbul
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi /ID# 239844, Istanbul
  - Ege University Medical Faculty /ID# 240139, Izmir
  - Necmettin Erbakan Universitesi /ID# 239848, Meram Konya

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M19-052